CLINICAL TRIAL: NCT01236209
Title: Stimulating Self Management in Patients With Fibromyalgia Through Web-based Situational Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: The Research Council of Norway (Other); St. Olavs Hospital (Other); Netherlands Instititute for Health Services Research (Other); Buskerud University College (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 182014/V50
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- web page (Active Comparator): Control group:
  Information web page with some mindfulness exercises
  Interventions: Other: Webpage
- Webpage and situational feedback (Experimental): Intervention group:
  have access to the same web-page with information about coping with pain and relaxation and are completing 3 diaries and receiving personalized feedback for 4 weeks at home through a smartphone.
  Interventions: Other: Webpage and situation feedback

INTERVENTIONS:
Other: Webpage — one arm having access to a webpage with information about coping with pain and relaxation exercises
  Other Names: Information web page with some mindfulness exercises
  Arms: web page
Other: Webpage and situation feedback — having access to the same web-page with information about coping with pain and relaxation relaxation and completing 3 diaries and receiving situational feedback for 4 weeks at home through a web enabled mobile phone.
  Other Names: Intervention group
  Arms: Webpage and situational feedback

SUMMARY:
The overall objective of this randomized controlled study (RCT) financed by the Norwegian Research Council (grant no. 182012/V50) is to establish the effectiveness of situational feedback to the self-management of fibromyalgia syndrome (FMS) using innovative means of patient-provider communication in a randomized controlled study (RCT). Thereby this project will contribute to the knowledge of treatment of patients with FMS. The effectiveness of the intervention will be expressed in terms of a) reduced pain, b) psychometric outcomes, c) quality of life, d) improved engagement in daily activities and e) prevented transition to chronic disability. We furthermore aim to 1) determine the effectiveness of providing regular situational feedback in enhancing self-management and, consequently 2) study the effectiveness of enhancing self-management in reducing pain and physical disability.

Self-management of chronic pain is increasingly seen as an important tool in providing adequate care to patients with FMS and other types of Chronic Non-malignant Pain. Enhancing the patient's self-management of her/his condition is thought to be effective in reducing pain and disability. However, sufficient empirical evidence to support this is yet unavailable. This may be due to the non-situational nature of many interventions studied so far: Patients are taught management skills in a clinical setting, and may not be able to successfully use these skills in daily care. Therefore, enhancing self-management of chronic pain, by providing immediate feedback that is directly related to patient's daily life ("situational" feedback) complementary to care-as usual, is thought to be more effective than conventional interventions in a clinical setting. This may even be even more effective when the patient receives quick response feedback using mobile communication technology, i.e. any place any time.

ELIGIBILITY:
Inclusion Criteria:

* Female, having wide spread pain like FMS (IPCS codes CD-10, 79.0 - coded) for at least three months ,> 18 years, able to understand Norwegian; able to use the webenabled mobile phone.

Exclusion Criteria:

* substantial psychological problems in need of treatment with intensive psychotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in catastrophizing cognitions | T1: At the start of in-house rehabilitation T2: At the end of in-house rehabilitation - begin situational feedback intervention T3: End of situational feedback intervention T4: 6 month after T1 T5: 12 months after T1
  PCS: Pain Catastrophizing Scale (Sullivan et al., 1995).

SECONDARY OUTCOMES:
Change in acceptance | T1: At the start of in-house rehabilitation T2: At the end of in-house rehabilitation - begin situational feedback intervention T3: End of situational feedback intervention T4: 6 month after T1 T5: 12 months after T1
  CPAQ: Chronic Pain Acceptance questionnaire (McCracken)

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Eide, PhD, Principal Investigator — Buskerud University College
Locations (1):
- Jeloy kurbad rehabilitation centre, Moss, Norway

REFERENCES:
- [Background] Nes AA, van Dulmen S, Wicksell R, Fors EA, Eide H. Analyzing Change Processes Resulting from a Smartphone Maintenance Intervention Based on Acceptance and Commitment Therapy for Women with Chronic Widespread Pain. Int J Behav Med. 2017 Apr;24(2):215-229. doi: 10.1007/s12529-016-9590-7. PMID 27541314
- [Background] Nes AA, Eide H, Kristjansdottir OB, van Dulmen S. Web-based, self-management enhancing interventions with e-diaries and personalized feedback for persons with chronic illness: a tale of three studies. Patient Educ Couns. 2013 Dec;93(3):451-8. doi: 10.1016/j.pec.2013.01.022. Epub 2013 Feb 21. PMID 23433735
- [Background] Smedslund G, Eide H, Kristjansdottir OB, Nes AA, Sexton H, Fors EA. Do weather changes influence pain levels in women with fibromyalgia, and can psychosocial variables moderate these influences? Int J Biometeorol. 2014 Sep;58(7):1451-7. doi: 10.1007/s00484-013-0747-7. Epub 2013 Oct 17. PMID 24132549
- [Derived] Kristjansdottir OB, Fors EA, Eide E, Finset A, Stensrud TL, van Dulmen S, Wigers SH, Eide H. A smartphone-based intervention with diaries and therapist feedback to reduce catastrophizing and increase functioning in women with chronic widespread pain. part 2: 11-month follow-up results of a randomized trial. J Med Internet Res. 2013 Mar 28;15(3):e72. doi: 10.2196/jmir.2442. PMID 23538392
- [Derived] Kristjansdottir OB, Fors EA, Eide E, Finset A, Stensrud TL, van Dulmen S, Wigers SH, Eide H. A smartphone-based intervention with diaries and therapist-feedback to reduce catastrophizing and increase functioning in women with chronic widespread pain: randomized controlled trial. J Med Internet Res. 2013 Jan 7;15(1):e5. doi: 10.2196/jmir.2249. PMID 23291270
- [Derived] Kristjansdottir OB, Fors EA, Eide E, Finset A, van Dulmen S, Wigers SH, Eide H. Written online situational feedback via mobile phone to support self-management of chronic widespread pain: a usability study of a Web-based intervention. BMC Musculoskelet Disord. 2011 Feb 25;12:51. doi: 10.1186/1471-2474-12-51. PMID 21352516